CLINICAL TRIAL: NCT03151109
Title: Glenoid Bone Grafting for Reverse Shoulder Arthroplasty: Clinical and Radiographic Outcomes
Brief Title: Glenoid Bone Grafting for RTSA: Clinical & Radiographic Outcomes
Acronym: EPBG
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 201507050
Record Dates: First submitted 2017-03-08; First posted 2017-05-12 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Osteo Arthritis Shoulders
Keywords: reverse total shoulder arthroplasty; glenoid bone loss
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT Scan — CT scan at minimum 1 year post op

SUMMARY:
This study will look at patient radiographic and functional outcomes who have or will undergo a reverse, extended peg, shoulder arthroplasty (replacement) that requires the use of glenoid bone grafting.

DETAILED DESCRIPTION:
Glenoid bone loss is a known issue with reverse shoulder implants and can lead to issues with implant fixation and stability over time. To address this issue an extended peg glenoid baseplate is used and area around plate is augmented with bone (auto or allo)graft material to encourage bony callous growth around the implant. This study is to look at this area of concern and determine if glenoid bone loss is occurring in the patients where these measures have been taken to deter its development.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients who have undergone a reverse shoulder arthroplasty with the an extended peg baseplate and structural bone graft (autograft humeral head or allograft femoral head).
2. Adult patients who are indicated for a long-pegged baseplate and glenoid bone grafting (autograft humeral head or allograft femoral head) as part of their reverse shoulder arthroplasty in our clinic,
3. bone graft is truly structural involving at least 50% of the glenoid baseplate
4. may be a primary or a revision surgery

Exclusion Criteria:

1. patients with missing baseline (preop) data,
2. patients who are unwilling to participate in a final follow-up evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with substantial glenoid bone loss in the context of severe glenohumeral arthrosis, advanced cuff tear arthropathy or those who have undergone prior shoulder arthroplasty and have or will undergo a reverse shoulder replacement with structural bone graft to address the problem.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Radiographic Outcome | minimum 1 year post op
  Evaluate Bone Graft Incorporation - review images to determine signs of humeral or glenoid radiolucency, radiographic loosening, fracture, notching, and graft incorporation versus resorption on CT and/or XRay images.

SECONDARY OUTCOMES:
Functional outcomes at year one | collected at 1 year post surgery
  Evaluate postoperative clinical outcome scores
Functional outcomes at year two | collected 2 years post surgery
  Evaluate postoperative clinical outcome scores

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Chamberlain, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frankle M, Levy JC, Pupello D, Siegal S, Saleem A, Mighell M, Vasey M. The reverse shoulder prosthesis for glenohumeral arthritis associated with severe rotator cuff deficiency. a minimum two-year follow-up study of sixty patients surgical technique. J Bone Joint Surg Am. 2006 Sep;88 Suppl 1 Pt 2:178-90. doi: 10.2106/JBJS.F.00123. PMID 16951091
- [Background] Naveed MA, Kitson J, Bunker TD. The Delta III reverse shoulder replacement for cuff tear arthropathy: a single-centre study of 50 consecutive procedures. J Bone Joint Surg Br. 2011 Jan;93(1):57-61. doi: 10.1302/0301-620X.93B1.24218. PMID 21196544
- [Background] Nolan BM, Ankerson E, Wiater JM. Reverse total shoulder arthroplasty improves function in cuff tear arthropathy. Clin Orthop Relat Res. 2011 Sep;469(9):2476-82. doi: 10.1007/s11999-010-1683-z. PMID 21116759
- [Background] Henninger HB, Barg A, Anderson AE, Bachus KN, Burks RT, Tashjian RZ. Effect of lateral offset center of rotation in reverse total shoulder arthroplasty: a biomechanical study. J Shoulder Elbow Surg. 2012 Sep;21(9):1128-35. doi: 10.1016/j.jse.2011.07.034. Epub 2011 Oct 29. PMID 22036546
- [Background] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838
- [Background] Hamada K, Fukuda H, Mikasa M, Kobayashi Y. Roentgenographic findings in massive rotator cuff tears. A long-term observation. Clin Orthop Relat Res. 1990 May;(254):92-6. PMID 2323152
- [Background] Antuna SA, Sperling JW, Cofield RH, Rowland CM. Glenoid revision surgery after total shoulder arthroplasty. J Shoulder Elbow Surg. 2001 May-Jun;10(3):217-24. doi: 10.1067/mse.2001.113961. PMID 11408901
- [Background] Sirveaux F, Favard L, Oudet D, Huquet D, Walch G, Mole D. Grammont inverted total shoulder arthroplasty in the treatment of glenohumeral osteoarthritis with massive rupture of the cuff. Results of a multicentre study of 80 shoulders. J Bone Joint Surg Br. 2004 Apr;86(3):388-95. doi: 10.1302/0301-620x.86b3.14024. PMID 15125127